CLINICAL TRIAL: NCT01456104
Title: Immune Responses to Autologous Langerhans-type Dendritic Cells Electroporated With mRNA Encoding a Tumor-associated Antigen in Patients With Malignancy: A Single-arm Phase I Trial in Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-229
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Melanoma
Keywords: vaccine; stage IIB; stage IIC; stage III; stage IV (MIa); Langerhans-type dendritic cells; Immune Responses; 10-229
MeSH Terms: conditions — Melanoma

ARMS (1):
- vaccine (Experimental): This is a single-arm phase I trial in patients with AJCC stage IIB, IIC, III, and IV (MIa) melanoma in which autologous human Langerhans-type dendritic cells (CD34+hematopoietic progenitor cell (HPC)-derived Langerhans cells, or LCs) will be electroporated with mRNA encoding full-length murine tyrosinase-related peptide 2 (TRP2). LCs will also be loaded with control antigens (HLA-A*0201-restricted flu matrix peptide).
  Interventions: Biological: Langerhans-type dendritic cells (a.k.a. Langerhans cells or LCs)

INTERVENTIONS:
Biological: Langerhans-type dendritic cells (a.k.a. Langerhans cells or LCs) — Patients will receive a total of 5 vaccinations, comprising a primary immunization followed by four boosters at 3 week intervals with a window of ± 4 days. Vaccines will be dosed at 10x106 LCs per vaccine x 5.

SUMMARY:
This study is being done to see if the investigators can help the immune system to work against melanoma.

A dendritic cell is another type of white blood cell. It has most, if not all, of the proteins needed to make T cells work to destroy cancer cells. However, dendritic cells do not normally have the cancer proteins on their surface. The challenge then is to combine the antigens with dendritic cells to make a vaccine. The investigators think that the body's T cells might then react against the tumor and help destroy it.

This study will see if altered dendritic cells will make T cells work against tumor cells. The dendritic cells will be made in a lab and will carry the antigens. These cells then will be injected under the skin.

In this study, the investigators are trying to help the body make a stronger immune response against the cancer. The patient will get the same kind of dendritic cell vaccine used in the earlier study, but with one major difference. The dendritic cells will contain messenger-RNA (mRNA). Cells use mRNA to make proteins. The mRNA will be put into dendritic cells by a laboratory method called electroporation. The mRNA is never given to the patient directly. This mRNA will help the dendritic cell make a tumor antigen like what the cancer expresses. The dendritic cell can then put this tumor antigen on its surface so that the body could make a stronger immune response against the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of melanoma, AJCC stage IIB, IIC, III, or IV (MIa), with histologic confirmation by the Department of Pathology at MSKCC.
* Patients must be HLA-A*0201 positive, based on high resolution DNA level typing.
* Expected survival of greater than 3 months.
* Karnofsky performance status of 70 or higher
* All patients should have undergone surgical treatment appropriate to their stage of disease
* Patients may not have received chemotherapy, immunotherapy, or radiation within a minimum of 28 days (minimum of 42 days for nitrosoureas or mitomycin) before participation in this protocol.

Exclusion Criteria:

* Pregnant or lactating women because of unknown risks to the fetus or infant.
* Patients requiring systemic corticosteroids or comparable exogenous immunosuppressive agent(s) (no exclusion for use of NSAIDs).
* Patients with a known immunodeficiency (e.g., infection with HTLV-1,2, HIV-1,2; etc.).
* Patients with coexisting autoimmune diseases, except vitiligo.
* Patients with baseline impairments of hematologic, hepatic, or renal function (CTCAE v4.0 > grade 1, ANC < 1500, hgb < 10.0 g/dl, plts < 75,000/ul, AST > 3x ULN, creatinine > 1.5xULN), all assessed within four weeks of study entry.
* Patients with organ allografts.
* Patients who are status post splenectomy or status post splenic irradiation.
* Patients with a history of documented pre-existing retinal/choroidal disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2011-10-17 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
safety | 1 year
  Toxicity will be graded according to standard NCI/CTEP toxicity criteria. This protocol will use the Common Terminology Criteria for Adverse Events (CTCAE) v4.0
toxicity | 1 year
  Toxicity will be graded according to standard NCI/CTEP toxicity criteria. This protocol will use the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Due to the nature of this treatment and the expected mild erythema and occasional pruritus, only grade 3-4 toxicities will be evaluated

SECONDARY OUTCOMES:
immunogenicity | 1 year
  For this study, the vaccine is considered promising if more than four out of the nine patients have an immunologic response (e.g., tetramer staining and intracellular cytokine secretion assays). Samples taken after vaccination will be considered positive for response if they are higher than the pre-vaccination values by at least two standard deviations. For each patient, the standard deviation of the background (calculated using triplicates) will be computed, and a positive will be defined as greater than two times this value.

CONTACTS AND LOCATIONS:
Overall Officials: James Young, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm